CLINICAL TRIAL: NCT00896246
Title: Scintigraphic Assessment of Gastrointestinal Transit Following Administration of Klean-Prep® (4L) or Moviprep® (2L) to Healthy Volunteers.
Brief Title: Scintigraphic Assessment Following Klean-Prep® or Moviprep®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Hans-Jürgen Gruss, Norgine Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRL994-01/2007 (GLO)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Gastric Emptying; Healthy
MeSH Terms: interventions — klean prep; MoviPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Klean-Prep® (Active Comparator): 1 x gelatin capsule containing not more than 1 MBq 111In radiolabelled ion exchange resin plus Klean-Prep® (4 L) containing 99mTc-DTPA administered as a divided dose.
  Interventions: Drug: Klean-Prep®
- Moviprep® (Experimental): 1 x gelatin capsule containing not more than 1 MBq 111In radiolabelled ion exchange resin plus Moviprep® (2 L) containing radiolabelled 99mTc-DTPA administered as a divided dose.
  Interventions: Drug: Moviprep®

INTERVENTIONS:
Drug: Klean-Prep® — Four litres of solution administered orally as a divided dose.
  Arms: Klean-Prep®
Drug: Moviprep® — Two litres of solution administered orally as a divided dose
  Arms: Moviprep®

SUMMARY:
This was a phase 1, open-label, randomized study, designed to assess the impact of Moviprep® or Klean-Prep® on gastrointestinal transit. It was performed in two parallel groups with Part A in two groups of four subjects preceding Part B, which was performed in two groups of 12 subjects. Subjects attended a pre-study medical within 28 days of dosing and a post-study medical 5-10 days after the final dose. Within both Part A and Part B, subjects were required to attend the clinical unit for 2 study periods. Part A consisted of a baseline period to determine individual reference times for gastrointestinal transit. Part B was the test period in which gastrointestinal transit following the administration of the test preparations was assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males;
2. Aged 18-65 years;
3. Body Mass Index of 18-35 kg/m2;
4. Must be willing and able to participate in the whole study and must provide written informed consent.

Exclusion Criteria:

1. Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months;
2. Subjects who have previously been enrolled in this study;
3. Subjects who have ever sought advice from or been referred to a GP or counsellor for abuse or misuse of alcohol, non medical drugs, medicinal drugs or other substance abuse e.g. solvents;
4. Subjects who admit to any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, LSD (d lysergic acid diethylamide) and intravenous amphetamines. Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have abstained from cannabis use for at least 3 months;
5. Positive drugs of abuse test result;
6. Regular alcohol consumption > 21 units per week (1 Unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine);
7. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening;
8. Radiation exposure from clinical trials, including that from the present study and from diagnostic x rays but excluding background radiation, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study;
9. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the PMI;
10. History of gastrointestinal surgery (with the exception of appendectomy unless it was performed within the previous 12 months);
11. History of clinically significant cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome;
12. Subjects with a hypersensitivity to any of the ingredients in either Moviprep® or Klean- Prep®;
13. Diarrhoea or constipation in the 7 days before the predicted first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day.
14. Subjects will be excluded from the study if they are considered by the PMI to be at risk of transmitting, through blood or other body fluids, the agents responsible for AIDS (Acquired Immunodeficiency Syndrome), other sexually transmitted disease or hepatitis. This will be assessed by the use of a question which requires that a potential subject decides whether he fulfills any category included on a reference card. If the answer is 'yes', the subject is excluded from the study;
15. Positive HBV, HCV or HIV results;
16. Subjects receiving prohibited medication as described in Section 7.4. Subjects must not stop taking a prescribed medication for the purpose of entering the study;
17. Subjects with a history of phenylketonuria or glucose-6-phosphate dehydrogenase deficiency;
18. Failure to satisfy the PMI of fitness to participate for any other reason.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To assess the impact of Moviprep® and Klean-Prep® on time of colonic transit of the contents of the colon in comparison to baseline | 2-4 days

SECONDARY OUTCOMES:
To assess the gastrointestinal transit of Moviprep® and Klean-Prep® in comparison to baseline | 2-4 days
To determine gastric emptying of Moviprep® and Klean-Prep® | 2-4 days
To collect information about stool weight, visual characteristics and distribution of the radiolabel | 2-4 days

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; Philip Evans, MB ChB MRCS, Principal Investigator — Pharmaceutical Profiles Ltd
Locations (1):
- Pharmaceutical Profiles Ltd, Nottingham, United Kingdom